CLINICAL TRIAL: NCT05592275
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of LY3540378 in Adults With Worsening Chronic Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: A Study of LY3540378 in Participants With Worsening Chronic Heart Failure With Preserved Ejection Fraction (HFpEF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: An interim was conducted and after review of available data, including efficacy evaluation of heart failure events, Lilly is terminating the study due to low likelihood of study success for this HFpEF patient population.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18473; J3E-MC-EZDB (Other: Eli Lilly and Company); 2023-505902-40-00 (Other: EU Trial Number)
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 25 mg LY3540378 (Experimental): Participants received 25 mg LY3540378 administered once weekly as subcutaneous (SC) injection for 26 weeks.
  Interventions: Drug: LY3540378
- 50 mg LY3540378 (Experimental): Participants received 50 mg LY3540378 administered once weekly as SC injection for 26 weeks.
  Interventions: Drug: LY3540378
- 100 mg LY3540378 (Experimental): Participants received 100 mg LY3540378 administered once weekly as SC injection for 26 weeks.
  Interventions: Drug: LY3540378
- Placebo (Placebo Comparator): Participants received placebo administered once weekly as SC injection for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3540378 — Administered SC
  Arms: 100 mg LY3540378; 25 mg LY3540378; 50 mg LY3540378
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of LY3540378 in adults with worsening heart failure with preserved ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* Experienced an index event, defined as a recent hospitalization for HF requiring ≥1 bolus doses of intravenous diuretics or an out- of- hospital encounter (for example, Emergency Room, clinic visit, infusion clinic, etc.) for HF requiring ≥1 bolus doses of intravenous diuretics.
* Documented LVEF of ≥50% within 12 months prior to screening; as measured by echocardiography, radionuclide ventriculography, invasive angiography, magnetic resonance imaging (MRI), or computerized tomograph (CT).
* Evidence of documentation of LVEF of ≥50% may also include participant medical records, discharge notes or a referral letter from the participant's physician or referring physician that details the participant's medical history.
* Had evidence of clinical HF syndrome consisting of hospitalization for worsening heart failure (WHF) with intravascular volume overload (the index event), as determined by the investigator, based on appropriate supportive documentation at randomization, and defined by ≥2 of the following:

  * dyspnea
  * jugular venous distention
  * pitting edema in lower extremities (>1+)
  * ascites
  * pulmonary congestion on chest X-ray
  * pulmonary rales AND participant received treatment with IV diuretics.

OR

* Treatment for an urgent visit outside of of being hospitalized with WHF and intravascular volume overload (the index visit) requiring treatment with IV diuretics (defined as ≥2 IV doses) such as in the outpatient setting/emergency room/observation unit/infusion clinic with a clinical response within the past 2 weeks prior to randomization. Urgent visit is defined as an unplanned visit for HF defined by ≥2 of the following:

  * dyspnea
  * jugular venous distention
  * pitting edema in lower extremities (>1+)
  * ascites
  * pulmonary rales on lung examination.
* NT-proBNP (>300 [sinus rhythm] or 600 pg/mL [atrial fibrillation or atrial flutter] OR BNP (>100 [sinus rhythm] or 200 pg/mL [atrial fibrillation or atrial flutter]) at screening.
* eGFR of >20 mL/min/1.73 m² at V1 (screening; determined by local laboratory), derived from serum creatinine values, age, and sex based on the CKD-EPI equation.

Exclusion Criteria

* Prior documentation of low ventricle ejection fraction (LVEF) ≤45% in the past 12 months.
* Have had acute coronary syndrome or percutaneous coronary intervention, coronary artery bypass graft, cardiac mechanical support implantation, within 3 months prior to V2. (randomization), - or any other cardiac surgery planned during the study.
* Have had left ventricular assist device (LVAD) or cardiac transplantation or have cardiac transplantation planned during the study.
* Have hypertrophic cardiomyopathy (obstructive or nonobstructive), restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, cardiac sarcoidosis, known amyloid cardiomyopathy, or inherited cardiomyopathy.
* Have a chronic pulmonary/lung disease (COPD), (pulmonary arterial hypertension, etc) as defined by chronic oxygen dependence. Night-time oxygen is not exclusionary.
* Uncorrected thyroid disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (137):
- United States (22):
  - Pima Heart, Tucson, Arizona
  - Valley Clinical Trials, Inc., Covina, California
  - Valley Clinical Trials, Inc., Northridge, California
  - University of California Irvine Medical Center, Orange, California
  - Pasadena Clinical Research, Pasadena, California
  - Velocity Clinical Research, Coastal Heart Medical Group, Santa Ana, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Infinite Clinical Research, Miami, Florida
  - South Florida Research Solutions - North Flamingo Road, Pembroke Pines, Florida
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Abington Memorial Hospital, Abington, Pennsylvania
  - PharmaTex Research, Amarillo, Texas
  - Baylor Scott & White Health-Advanced Heart and Lung Disease, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - West Houston Area Clinical Trial Consultants, Houston, Texas
  - Texas Institute of Cardiology, PA, McKinney, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Argentina (15):
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Investigaciones Medicas Imoba Srl, Balvanera, Buenos Aires F.D.
  - Sanatorio Anchorena Recoleta, Buenos Aires, Buenos Aires F.D.
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Sanatorio San Martin, Venado Tuerto, Santa Fe Province
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán, Tucumán Province
  - CEMEDIC, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares, Santa Fe
- Brazil (15):
  - Centro de Pesquisa Silvestre Santé, Rio Branco, Acre
  - Universidade Federal de Goias, Goiânia, Goiás
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR, Curitiba, Paraná
  - Centro de Pesquisa Clinica do Coracao, Acaraju, Sergipe
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Instituto de Pesquisa clinica de Campinas, Campinas, São Paulo
  - Instituto Do Coracao De Marilia, Marília, São Paulo
  - CAPED Centro Avancado Pesquisa e Diagnostica, Ribeirão Preto, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - Hospital Santa Paula, São Paulo, São Paulo
  - Incor - Instituto do Coracao, São Paulo, São Paulo
  - Instituto de Molestias Cardiovasculares de Tatui, Tatuí, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
  - Hospital São Lucas de Copacabana, Rio de Janeiro
  - Instituto D'Or Pesquisa e Ensino, Rio de Janeiro
- Canada (9):
  - SMH Cardiology Clinical Trials, Surrey, British Columbia
  - Private Practice - Dr. Saul Vizel, Cambridge, Ontario
  - PACE Cardiology, Newmarket, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - Heart Health Institute - Scarborough Office, Scarborough Village, Ontario
  - Medicus MFC Research Clinic, Toronto, Ontario
  - CPS Research, Waterloo, Ontario
  - Centre Hospitalier Universite de Sherbrooke - Hôtel-Dieu Hospital, Sherbrooke, Quebec
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni Nemocnice u sv. Anny v Brne, Brno, South Moravian
  - Vseobecna fakultni nemocnice v Praze, Prague
- Hungary (6):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Medifarma 98 Kft, Nyíregyháza, Nyíregyháza
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa, Pest County
  - Belvárosi Egészségház, Zalaegerszeg, Zala County
  - Dél-Pesti Centrumkórház, Budapest
  - Semmelweis University, Budapest
- Israel (4):
  - Yitzhak Shamir Medical Center, Ẕerifin, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Japan (19):
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Saiseikai Futsukaichi Hospital, Chikushino-shi, Fukuoka
  - Nakamura Cardiovascular Clinic, Itoshima, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Takasaki General Medical Centar, Takasaki, Gunma
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokohama Minami Kyosai Hospital, Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Ome Medical Center, Ōme, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Harasanshin Hospital, Fukuoka
  - Rakuwakai Otowa Hospital, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Sakurabashi Watanabe Advanced Healthcare Hospital, Osaka
  - Yodogawa Christian Hospital, Osaka
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research, Osaka
  - Toyama Prefectural Central Hospital, Toyama
- Poland (14):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - INTERCOR, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Private Practice - Dr. Ewa Mirek Bryniarska, Krakow, Lesser Poland Voivodeship
  - MEDICOME Centrum Badań Klinicznych Oświęcimskie, Oświęcim, Lesser Poland Voivodeship
  - 1 Wojskowy Szpital Kliniczny w Lublinie, Lublin, Lublin Voivodeship
  - CenterMed Lublin NZOZ, Lublin, Lublin Voivodeship
  - Balsam Medica, Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl, Podkarpackie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok, Podlaskie Voivodeship
  - KLIMED Marek Klimkiewicz, Bialystok, Podlaskie Voivodeship
  - SPZOZ Uniwersytecki Szpital Kliniczny Im. Wojskowej Akademii Medycznej UM W Łodzi Centralny Szpital Wetera -T, Lodz, Łódź Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship
  - IRMED Osrodek Badan Klinicznych, Piotrkow Trybunalski, Łódź Voivodeship
  - Provita Profamilia, Piotrkow Trybunalski, Łódź Voivodeship
- Spain (12):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital de Denia Marina Salud, Denia, Alicante
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen de Valme, Seville, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [Barcelona]
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Hospital San Juan de la Cruz, Úbeda, Jaén
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Murcia, Región de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario 12 de Octubre, Madrid
- Turkey (Türkiye) (10):
  - Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi, Yıldırım, Bursa
  - Eskisehir Osmangazi University, Eskişehir, Eskişehir
  - Ege Universitesi Hastanesi, Bornova, İzmir
  - Kocaeli Üniversitesi, İzmit, Kocaeli
  - Afyon Kocatepe Üniversitesi Tıp Fakültesi, Afyonkarahisar
  - Ankara Etlik City Hospital, Ankara
  - Trakya University Medical Faculty Hospital, Edirne
  - T.C. Sağlık Bakanlığı İzmir Tepecik Eğitim ve Araştırma Hast, Izmir
  - Dokuz Eylul Universitesi Hastanesi, Izmir
  - Mersin University, Mersin
- United Kingdom (8):
  - Wycombe General Hospital, High Wycombe, Buckinghamshire
  - Raigmore Hospital, Inverness, Highland
  - Northwick Park Hospital, Harrow, London, City of
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - West Middlesex University Hospital, Isleworth
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Wythenshawe Hospital, Manchester
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Borlaug BA, Testani JM, Petrie MC, Wang Z, Cunningham J, Adams KF Jr, Amir O, Belohlavek J, Bocchi E, Freitas A Jr, Hominal M, Kadokami T, Merkely B, Miller CA, Nunez J, Verma S, Yilmaz MB, Oru E, Sam F. Effects of volenrelaxin in worsening heart failure with preserved ejection fraction: a phase 2 randomized trial. Nat Med. 2025 Nov;31(11):3853-3861. doi: 10.1038/s41591-025-03939-6. Epub 2025 Aug 31. PMID 40887551
- See also: A Study of LY3540378 in Participants With Worsening Chronic Heart Failure With Preserved Ejection Fraction (HFpEF) — https://trials.lilly.com/en-US/trial/366076

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Started | 79 | 83 | 81 | 89
Received at Least One Dose of Study Drug | 79 | 83 | 81 | 88
Completed | 45 | 48 | 43 | 46
Not Completed | 34 | 35 | 38 | 43
Not completed — Study Terminated by Sponsor | 17 | 22 | 21 | 27
Not completed — Site Terminated by Sponsor | 6 | 6 | 7 | 5
Not completed — Withdrawal by Subject | 3 | 2 | 6 | 3
Not completed — Death | 3 | 2 | 3 | 2
Not completed — Assigned Treatment by Mistake | 1 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 1 | 0 | 0 | 0
Not completed — Did not Follow Schedule of Activities by Uploading Echocardiograms Within Time | 1 | 0 | 0 | 0
Not completed — pro B-type Natriuretic Peptide was not Collected on Time | 1 | 0 | 0 | 0
Not completed — Sponsor Decision to Discontinue the Participant | 0 | 0 | 0 | 1
Not completed — Participant Refused to Participant in Study | 0 | 0 | 0 | 1
Not completed — Participant is Travelling | 0 | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 25 mg LY3540378: Participants received 25 mg LY3540378 administered once weekly as SC injection for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo | Total
Number analyzed (Participants) | 79 | 83 | 81 | 89 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.10 (10.08) | 74.70 (8.14) | 72.40 (9.69) | 74.60 (9.07) | 74.00 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 44 | 29 | 164
  Male | 33 | 38 | 37 | 60 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 39 | 34 | 37 | 151
  Not Hispanic or Latino | 37 | 44 | 45 | 52 | 178
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 3 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 8 | 3 | 18
  White | 72 | 74 | 68 | 79 | 293
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Argentina | 16 | 23 | 11 | 15 | 65
  Brazil | 17 | 9 | 19 | 17 | 62
  Canada | 2 | 4 | 0 | 3 | 9
  Hungary | 8 | 11 | 12 | 14 | 45
  Israel | 1 | 1 | 1 | 1 | 4
  Japan | 2 | 2 | 3 | 7 | 14
  Poland | 15 | 14 | 17 | 14 | 60
  Spain | 15 | 13 | 8 | 14 | 50
  United Kingdom | 0 | 2 | 2 | 1 | 5
  United States | 3 | 4 | 8 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Atrial Reservoir Strain (LARS) at Week 26
Description: Results are estimated using least squares (LS) mean from the mixed model repeated measures (MMRM) model: Change from baseline = Baseline + Strata + Gender + Treatment + Time + Treatment*Time + Baseline*Treatment.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline value at the specified time point for this outcome.
Measure: Least Squares Mean (Standard Error); unit: percentage strain
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 32 | 37 | 31 | 38
percentage strain | 1.924 (1.000) | -0.643 (0.926) | -1.048 (1.008) | -1.930 (0.931)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0058, Mixed Models Analysis; LS Mean Difference = 3.853, 95% CI 2-sided [1.14 to 6.57], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.3321, Mixed Models Analysis; LS Mean Difference = 1.286, 95% CI 2-sided [-1.33 to 3.90], Standard Error of Mean 1.32
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.5211, Mixed Models Analysis; LS Mean Difference = 0.881, 95% CI 2-sided [-1.83 to 3.59], Standard Error of Mean 1.37

2. Secondary Outcome: Change From Baseline in Left Atrial Reservoir Strain (LARS) at Week 12
Description: Results are estimated using LS mean from the MMRM model: Change from baseline = Baseline + Strata + Gender + Treatment + Time + Treatment*Time + Baseline*Treatment.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage strain
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 40 | 44 | 41 | 45
percentage strain | 0.250 (1.124) | -0.135 (1.078) | 1.313 (1.121) | -0.951 (1.061)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.4400, Mixed Models Analysis; LS Mean Difference = 1.201, 95% CI 2-sided [-1.86 to 4.27], Standard Error of Mean 1.55
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.5913, Mixed Models Analysis; LS Mean Difference = 0.816, 95% CI 2-sided [-2.18 to 3.81], Standard Error of Mean 1.52
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.1446, Mixed Models Analysis; LS Mean Difference = 2.265, 95% CI 2-sided [-0.79 to 5.31], Standard Error of Mean 1.54

3. Secondary Outcome: Change From Baseline in Log-transformed N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanogram per liter (ng/L)
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 50 | 55 | 47 | 58
nanogram per liter (ng/L) | 0.159 (0.081) | -0.092 (0.080) | 0.016 (0.084) | -0.112 (0.076)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0153, Mixed Models Analysis; LS Mean Difference = 0.272, 95% CI 2-sided [0.05 to 0.49], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.8509, Mixed Models Analysis; LS Mean Difference = 0.021, 95% CI 2-sided [-0.20 to 0.24], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.2558, Mixed Models Analysis; LS Mean Difference = 0.129, 95% CI 2-sided [-0.09 to 0.35], Standard Error of Mean 0.11

4. Secondary Outcome: Change From Baseline in Log-transformed N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) at Week 26
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanogram per liter (ng/L)
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 39 | 43 | 36 | 44
nanogram per liter (ng/L) | 0.095 (0.092) | -0.207 (0.088) | 0.010 (0.095) | -0.260 (0.086)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0050, Mixed Models Analysis; LS Mean Difference = 0.355, 95% CI 2-sided [0.11 to 0.60], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.6670, Mixed Models Analysis; LS Mean Difference = 0.053, 95% CI 2-sided [-0.19 to 0.30], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0350, Mixed Models Analysis; LS Mean Difference = 0.270, 95% CI 2-sided [0.02 to 0.52], Standard Error of Mean 0.13

5. Secondary Outcome: Change From Baseline in Left Atrial End-Diastolic Volume Index (LAEDVI) at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millilitres per square metre (mL/m²)
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 41 | 45 | 43 | 47
millilitres per square metre (mL/m²) | 0.921 (1.295) | 2.349 (1.249) | 0.899 (1.266) | 1.155 (1.205)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.8952, Mixed Models Analysis; LS Mean Difference = -0.235, 95% CI 2-sided [-3.74 to 3.27], Standard Error of Mean 1.78
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.4946, Mixed Models Analysis; LS Mean Difference = 1.193, 95% CI 2-sided [-2.25 to 4.63], Standard Error of Mean 1.74
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.8840, Mixed Models Analysis; LS Mean Difference = -0.256, 95% CI 2-sided [-3.72 to 3.21], Standard Error of Mean 1.75

6. Secondary Outcome: Change From Baseline in Left Atrial End-Diastolic Volume Index (LAEDVI) at Week 26
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/m²
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 33 | 38 | 32 | 38
mL/m² | -0.300 (1.416) | 2.978 (1.354) | 0.433 (1.425) | -1.388 (1.324)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.5763, Mixed Models Analysis; LS Mean Difference = 1.088, 95% CI 2-sided [-2.75 to 4.93], Standard Error of Mean 1.94
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0233, Mixed Models Analysis; LS Mean Difference = 4.366, 95% CI 2-sided [0.60 to 8.13], Standard Error of Mean 1.91
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.3504, Mixed Models Analysis; LS Mean Difference = 1.821, 95% CI 2-sided [-2.02 to 5.66], Standard Error of Mean 1.94

7. Secondary Outcome: Change From Baseline Left Atrial End-Systolic Volume Index (LAESVI) at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/m²
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 41 | 45 | 43 | 47
mL/m² | 4.893 (1.456) | 3.671 (1.412) | 3.637 (1.435) | 2.662 (1.364)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.2675, Mixed Models Analysis; LS Mean Difference = 2.231, 95% CI 2-sided [-1.73 to 6.19], Standard Error of Mean 2.01
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.6097, Mixed Models Analysis; LS Mean Difference = 1.009, 95% CI 2-sided [-2.89 to 4.90], Standard Error of Mean 1.97
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.6244, Mixed Models Analysis; LS Mean Difference = 0.975, 95% CI 2-sided [-2.95 to 4.90], Standard Error of Mean 1.99

8. Secondary Outcome: Change From Baseline Left Atrial End-Systolic Volume Index (LAESVI) at Week 26
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/m²
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 33 | 38 | 32 | 38
mL/m² | 2.922 (1.693) | 6.371 (1.617) | 2.455 (1.711) | 0.967 (1.591)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.4025, Mixed Models Analysis; LS Mean Difference = 1.955, 95% CI 2-sided [-2.65 to 6.56], Standard Error of Mean 2.33
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0191, Mixed Models Analysis; LS Mean Difference = 5.404, 95% CI 2-sided [0.90 to 9.91], Standard Error of Mean 2.28
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.5248, Mixed Models Analysis; LS Mean Difference = 1.488, 95% CI 2-sided [-3.13 to 6.10], Standard Error of Mean 2.34

9. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 12
Description: Results are estimated using LS mean from the MMRM model: Change from baseline = Baseline + Strata + Gender + Treatment + Time + Treatment*Time + Baseline*Treatment.
  The unit of measure for this outcome is millilitres per minute per 1.73 square metres (mL/min/1.73 m²)
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m²
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 51 | 54 | 47 | 60
mL/min/1.73 m² | 5.507 (1.394) | 6.303 (1.352) | 3.483 (1.425) | 0.439 (1.297)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0086, Mixed Models Analysis; LS Mean Difference = 5.067, 95% CI 2-sided [1.30 to 8.84], Standard Error of Mean 1.91
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0020, Mixed Models Analysis; LS Mean Difference = 5.863, 95% CI 2-sided [2.16 to 9.57], Standard Error of Mean 1.88
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.1160, Mixed Models Analysis; LS Mean Difference = 3.044, 95% CI 2-sided [-0.76 to 6.84], Standard Error of Mean 1.93

10. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 26
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m²
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 38 | 44 | 37 | 45
mL/min/1.73 m² | 4.848 (1.888) | 4.273 (1.788) | 3.048 (1.915) | 1.787 (1.743)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.2360, Mixed Models Analysis; LS Mean Difference = 3.061, 95% CI 2-sided [-2.02 to 8.14], Standard Error of Mean 2.58
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.3216, Mixed Models Analysis; LS Mean Difference = 2.486, 95% CI 2-sided [-2.45 to 7.42], Standard Error of Mean 2.50
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.6269, Mixed Models Analysis; LS Mean Difference = 1.261, 95% CI 2-sided [-3.85 to 6.37], Standard Error of Mean 2.59

11. Secondary Outcome: Change From Baseline in Log-transformed Serum Creatinine at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 51 | 55 | 47 | 62
milligram per deciliter (mg/dL) | -0.163 (0.027) | -0.112 (0.026) | -0.072 (0.028) | 0.015 (0.025)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.178, 95% CI 2-sided [-0.25 to -0.11], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0005, Mixed Models Analysis; LS Mean Difference = -0.127, 95% CI 2-sided [-0.20 to -0.06], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0219, Mixed Models Analysis; LS Mean Difference = -0.087, 95% CI 2-sided [-0.16 to -0.01], Standard Error of Mean 0.04

12. Secondary Outcome: Change From Baseline in Log-transformed Serum Creatinine at Week 26
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 39 | 44 | 37 | 45
milligram per deciliter (mg/dL) | -0.125 (0.030) | -0.083 (0.028) | -0.066 (0.030) | -0.007 (0.027)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0038, Mixed Models Analysis; LS Mean Difference = -0.117, 95% CI 2-sided [-0.20 to -0.04], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0558, Mixed Models Analysis; LS Mean Difference = -0.075, 95% CI 2-sided [-0.15 to 0.00], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.1496, Mixed Models Analysis; LS Mean Difference = -0.059, 95% CI 2-sided [-0.14 to 0.02], Standard Error of Mean 0.04

13. Secondary Outcome: Change From Baseline in Log-transformed Cystatin-C at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 52 | 55 | 47 | 60
milligram per liter (mg/L) | -0.064 (0.022) | -0.060 (0.021) | -0.040 (0.023) | -0.007 (0.020)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0569, Mixed Models Analysis; LS Mean Difference = -0.057, 95% CI 2-sided [-0.12 to 0.00], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.0683, Mixed Models Analysis; LS Mean Difference = -0.054, 95% CI 2-sided [-0.11 to 0.00], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.2738, Mixed Models Analysis; LS Mean Difference = -0.033, 95% CI 2-sided [-0.09 to 0.03], Standard Error of Mean 0.03

14. Secondary Outcome: Change From Baseline in Log-transformed Cystatin-C at Week 26
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
Number analyzed (Participants) | 38 | 44 | 37 | 45
mg/L | -0.058 (0.023) | -0.037 (0.025) | -0.036 (0.024) | -0.040 (0.026)
Statistical Analysis 1: Comparison: 25 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.5320, Mixed Models Analysis; LS Mean Difference = 0.021, 95% CI 2-sided [-0.05 to 0.09], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: 50 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.4974, Mixed Models Analysis; LS Mean Difference = 0.023, 95% CI 2-sided [-0.04 to 0.09], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: 100 mg LY3540378 vs Placebo; Test type: Superiority; p = 0.6016, Mixed Models Analysis; LS Mean Difference = 0.018, 95% CI 2-sided [-0.05 to 0.09], Standard Error of Mean 0.03

ADVERSE EVENTS:
Time Frame: Baseline up to Week 30
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 25 mg LY3540378 | 50 mg LY3540378 | 100 mg LY3540378 | Placebo
All-Cause Mortality (participants affected / at risk) | 3/79 | 2/83 | 3/81 | 2/88
Serious Adverse Events (participants affected / at risk) | 19/79 | 26/83 | 20/81 | 15/88
Other Adverse Events (participants affected / at risk) | 50/79 | 57/83 | 46/81 | 55/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 25 mg LY3540378 (N=79) | 50 mg LY3540378 (N=83) | 100 mg LY3540378 (N=81) | Placebo (N=88)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Cardiac failure (Cardiac disorders) | 4 (5) | 9 (12) | 5 (10) | 3 (5)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal haemorrhage (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial atrophy (Reproductive system and breast disorders) | 0/46 (0) | 1/45 (1) | 0/44 (0) | 0/29 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/46 (0) | 1/45 (1) | 0/44 (0) | 0/29 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 25 mg LY3540378 (N=79) | 50 mg LY3540378 (N=83) | 100 mg LY3540378 (N=81) | Placebo (N=88)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 6 (6) | 5 (5) | 3 (3)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic cyst (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 6 (6) | 5 (6) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 8 (14) | 11 (14) | 7 (9) | 6 (6)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Heart alternation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye haematoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Oral mucosal eruption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 0 (0) | 3 (4) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 2 (19) | 3 (5) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 5 (6) | 5 (5) | 1 (1) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 5 (6) | 2 (2) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (3) | 4 (5) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 3 (3) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (4) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (4) | 3 (4) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (4) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Inflammatory marker increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Volume blood increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calcium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food aversion (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 2 (3) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (2) | 2 (2)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/33 (0) | 0/38 (0) | 0/37 (0) | 1/59 (1)
Tumour of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 4 (5) | 1 (1)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Discouragement (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Albuminuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (3) | 2 (2)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/33 (0) | 1/38 (1) | 0/37 (0) | 0/59 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2/33 (2) | 1/38 (1) | 0/37 (0) | 0/59 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/46 (0) | 0/45 (0) | 1/44 (1) | 0/29 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/46 (0) | 1/45 (1) | 0/44 (0) | 1/29 (1)
Varicocele (Reproductive system and breast disorders) | 0/33 (0) | 1/38 (1) | 0/37 (0) | 0/59 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/46 (0) | 0/45 (0) | 1/44 (1) | 0/29 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 3 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 2 (4) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardioversion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal pessary removal (Surgical and medical procedures) | 0/46 (0) | 0/45 (0) | 1/44 (1) | 0/29 (0)
Vocal cord polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Hypotension (Vascular disorders) | 3 (3) | 5 (7) | 5 (8) | 6 (7)
Orthostatic hypotension (Vascular disorders) | 2 (3) | 1 (8) | 4 (5) | 1 (3)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT05592275/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT05592275/SAP_001.pdf